CLINICAL TRIAL: NCT04140006
Title: Evaluation of Topical Application of Alendronate Sodium In-situ Gel and Recombinant Human Bone Morphogenic Protein 2 on Dental Implant Stability and Crestal Bone Level: A Randomized Controlled Clinical Study
Brief Title: Efficacy of Antiresorptive and Bone Forming Material on Dental Implants
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Dhuha A. Al-assaf, Principal investigator, University of Baghdad
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 034118
Record Dates: First submitted 2019-06-26; First posted 2019-10-25 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Partial Edentulism
MeSH Terms: interventions — Bone Morphogenetic Protein 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Alendronate Gel (ALN) (Active Comparator): After preparation, 0.05 ml of the gel containing 100 µg of ALN will be injected in the osteotomy site immediately before fixture insertion (20 fixtures)
  Interventions: Drug: ALN Gel
- Bone Morphogenic Protein Gel (BMP) (Active Comparator): After preparation, 0.05 ml of the gel containing 100 µg of BMP will be injected in the osteotomy site immediately before fixture insertion (20 fixtures)
  Interventions: Drug: BMP Gel
- Mixture Gel of ALN and BMP (Active Comparator): After preparation, 0.05 ml of mixture gel containing 50 µg of ALN and 50 µg of BMP will be injected in the osteotomy site immediately before fixture insertion (20 fixtures)
  Interventions: Drug: Mixed Gel
- Control (Sham Comparator): After preparation, the fixture will be inserted without topical application of any medication (20 fixtures)
  Interventions: Drug: Control

INTERVENTIONS:
Drug: ALN Gel — Flapped surgery for insertion of dental implant with topical application of ALN gel
  Other Names: Alendronate Sodium trihydrate, m.w 325.12, Pharmaceutical Secondary standard, PHR 1599
  Arms: Alendronate Gel (ALN)
Drug: BMP Gel — Flapped surgery for insertion of dental implant with topical application of BMP gel
  Other Names: CowellBMP, recombinant human bone morphogenic protein type 2, rhBMP2
  Arms: Bone Morphogenic Protein Gel (BMP)
Drug: Mixed Gel — Flapped surgery for insertion of dental implant with topical application of mixed gel of ALN and BMP
  Other Names: Mixture of Alendronate Sodium trihydrate, m.w 325.12, Pharmaceutical Secondary standard, PHR 1599, and CowellBMP, recombinant human bone morphogenic protein type 2, rhBMP2
  Arms: Mixture Gel of ALN and BMP
Drug: Control — Flapped surgery for insertion of dental implant without topical application of any gel
  Other Names: No treatment
  Arms: Control

SUMMARY:
Insertion of a metal implant is considered one of the most common surgeries for fracture treatment, joint replacement, and dental implants. The success rate of these implants depends on their fixation which is in turn related primarily on the strength of the bone holding them. Studies evaluating the influence of local application of antiresorptive drugs, like bisphosphonates, on implanted endoprostheses whether orthopedic or dental is increasing annually with more and more experimental studies as well as clinical trials worldwide. On the other hand implants that release medications that enhance bone formation will lead to improved implant fixation and success. The objective of this study was to evaluate the effect of topical application of alendronate sodium gel and recombinant human bone morphogenic protein 2 on dental implant stability and crestal bone level.

DETAILED DESCRIPTION:
Bisphosphonates (BPs), which are so called because they have two phosphonate (PO3) groups, are structurally similar to natural pyrophosphate (PP), a normal product of human metabolism that has a calcium chelating property. They are used to treat bone metastases, osteoporosis, Paget's disease, and other skeletal disorders.

During bone remodeling, osteoclast bone resorptive action is impeded by BPs which are released into the resorption lacunae. These cells take up BPs from resorption lacunae and the BPs then trigger the osteoclasts to undergo apoptosis. It has been found that an adjunct treatment of implant site with BPs solution might be beneficial to initial osseointegration of immediately or delayed loaded dental implants without interfering significantly with peri-implant bone remodeling over time.

Oral or intravenous administrations are the classical BPs treatment modalities with many studies show their positive effect on peri-implant bone. More efficient delivery systems to the target sites have been investigated to minimize BPs side effects and alter their biodistribution in order to improve their bioavailability; one of those new systems is topical application. Topical application of BPs enhances osseointegration, promote implant-bone contact and increase the amount of bone peripheral to dental implants. Minimal amounts of bisphosphonates was found to improve early implant fixation and to be less prone to cause osteonecrosis of the jaw, this might lead to new possibilities for orthopedic surgery in osteoporotic bones and for dental implants with a smaller risk of such complication in comparison with systemic treatment.

In order to maximize anabolism and minimize catabolism, new coating strategies have been evolved to enhanced bone formation onto the implant surface which is more desired than only reduce bone resorption around it. So to improve implant osseointegration, a dedicated drug-loading ability to locally target bone disorders has been developed to combine antiresorptive and anabolic agents, such as bone morphogenic protein, which for instance and in osteoporotic bone, will improve bone healing process.

With a view to diminishing the side effects caused by the systemic use of BPs, such as oesophagitis and osteonecrosis of the jaw, and to maximize anabolism and minimize catabolism, recent studies have sought alternative systems for local delivery of these agents with or without bone forming agent, either by means of immobilizing on the implant surface (coating or immersion in BPs solution), or by applying the drug directly to the surgical site before implant insertion either as an irrigant or gel.

ELIGIBILITY:
Inclusion criteria Otherwise healthy patients over 18 years or with systemic diseases that do not interfere with bone healing Having single or multiple missing teeth in maxilla and/or mandible Having an alveolar ridge of sufficient vertical and horizontal dimensions and considered straightforward cases according to SAC classification

Exclusion criteria Patients with active or chronic infection or inflammation in the implant zone History of radiotherapy to the head and neck Past or current treatment with oral/intramuscular/intravenous bisphosphonates or other drugs altering bone metabolism Heavy smokers or with sever periodontitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Implant stability | 8 weeks
  Mean implant stability between different comparators following implants insertion by using resonance frequency analysis scaled from 1 to 100
Implant stability | 12 weeks post surgery
  Mean implant stability between different comparators following implants insertion by using resonance frequency analysis scaled from 1 to 100
Implant stability | 12 weeks post loading
  Mean implant stability between different comparators following implants loading by using resonance frequency analysis scaled from 1 to 100
Crestal bone level | 12 weeks post surgery
  Mean crestal bone level between different comparators following implants insertion by using cone beam computerized tomography measured from the first bone implant contact by millimeters
Crestal bone level | 12 weeks post loading
  Mean crestal bone level between different comparators following implants loading by using cone beam computerized tomography measured from the first bone implant contact by millimeters

SECONDARY OUTCOMES:
Bone density around dental implant | 12 weeks post surgery
  Mean difference in bone density around dental implants between different comparators following implants insertion by using cone beam computerized tomography with hounsfield unit
Bone density around dental implant | 12 weeks post loading
  Mean difference in bone density around dental implants between different comparators following implants loading by using cone beam computerized tomography with hounsfield unit

CONTACTS AND LOCATIONS:
Overall Officials: Salwan Y Bede, Principal Investigator — University of Baghdad
Locations (1):
- College of dentistry, University of Baghdad, Baghdad, Bab-Almoadham, Iraq

IPD SHARING:
Plan to Share IPD: No